CLINICAL TRIAL: NCT04723615
Title: Evaluation of Turkish Validity, Reliability and Practicality of Örebro Musculoskeletal System Screening Questionnaire-12
Brief Title: Orebro Musculoskeletal Screening Questionnaire-12
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2020/469
Record Dates: First submitted 2021-01-17; First posted 2021-01-26 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Musculoskeletal Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Orebro Musculoskeletal Screening Questionnaire-12 — It is a 12-item self-report questionnaire that aims to estimate the severity of the problem, functional impairment, reporting status, cost and recovery time in musculoskeletal problems.
Other: Visual Analog Scale — A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
Other: The Tampa Scale of Kinesiophobia — The Tampa Scale of Kinesiophobia that was developed in 1990 is a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain.
Other: Short Form-12 (SF-12) — The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.

SUMMARY:
The research is a study with methodological design. The validity, reliability and practicality of the Örebro Musculoskeletal System Screening Questionnaire-12 will be investigated. In this context, a questionnaire will be applied to the participants to take part in the study after the translation process is completed.

DETAILED DESCRIPTION:
Musculoskeletal disorders are quite common in developed and developing countries. Musculoskeletal disorders cause economic burdens in the individual and social field. In addition, getting reports is one of the main causes of reduced productivity and work disability. Therefore, inexpensive and easily applicable screening questionnaires are needed to determine the patient population with high risk musculoskeletal disorders. The Örebro Musculoskeletal Screening Questionnaire is a practical questionnaire that can evaluate musculoskeletal disorders and is tailored to the WHO-ICF themes. For this reason, the aim of the study is to translate the Örebro Musculoskeletal System Survey-12 into Turkish intercultural translation and to investigate the construct validity, reliability and practicality.

ELIGIBILITY:
Inclusion Criteria:

* Having any musculoskeletal problems (spine, upper or lower extremities)
* Being in the age range of 18-65

Exclusion Criteria:

* Pregnancy
* Having of red flag signs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be contacted via Google forms after the entire translation process of the questionnaire is completed. Participants will be 18-65 years and have any musculoskeletal problems (spine, upper or lower extremities).
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-12-18 (Estimated); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Orebro Musculoskeletal Screening Questionnaire-12 | 10 minutes
  It is a 12-item self-report questionnaire that aims to estimate a wide range of outcomes (severity of the problem, functional impairment, reporting status, cost and recovery time) in patients with acute and subacute work injury presenting with musculoskeletal pain involving the spine, upper and lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Derived] Tasvuran Horata E, Demir P, Yagci G, Erel S, Eken F, Gabel CP. The validity and reliability of the Turkish version of the 12-item Orebro musculoskeletal screening questionnaire (OMSQ-12-TR). Disabil Rehabil. 2023 Dec;45(25):4288-4295. doi: 10.1080/09638288.2022.2089918. Epub 2022 Jun 25. PMID 35758151